CLINICAL TRIAL: NCT00710320
Title: Temperature Changes During Induction of General Anesthesia in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Mohanad Shukry/MD, University of Oklahoma Health Siences Center/Pediatric Anesthesiology
Other Study IDs: IRB No 14004
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Hypothermia
Keywords: Children core temperature,; Pediatric surgery,; Anesthesia induction
MeSH Terms: conditions — Hypothermia | interventions — Temperature; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cover and Uncover: Procedure/Surgery
  Interventions: Procedure: Covered and uncovered anesthesia induction

INTERVENTIONS:
Procedure: Covered and uncovered anesthesia induction — We hypothesize that the core temperatures of:
  1. the covered group during induction of general anesthesia will be greater by 0.5ºC than the uncovered group during induction of general anesthesia.
  2. both groups, covered and uncovered, will be equal during surgery and post-operatively. In other words, due to the active warming procedures during surgery and post-operatively in the PICU, core temperatures of the uncovered group will catch up to the covered group.
  Other Names: Temperature; Pediatric; Urology; Anesthesia

SUMMARY:
We aim that uncovering patients during induction of general anesthesia does not decrease core body temperature in pediatric patients.

DETAILED DESCRIPTION:
Some anesthesiologists cover the pediatric patient with a blanket during the induction of general anesthesia, while others do not. Complaints have been raised by pediatric surgeons that if a pediatric patient is not covered during induction of general anesthesia, the child's core body temperature will be lower than normal following surgery and in the recovery room.

Children are at risk of significant heat loss in the operating room due to multiple factors, such as, exposure to cold temperatures, decrease in metabolism following induction of general anesthesia, increased surface-area-to-volume ratio, and through considerable respiratory heat loss.1

A decrease in temperature of 0.5ºC to 1.5ºC can occur during induction of general anesthesia in pediatric patients2. The use of heating blankets and warmers may increase temperature or result in a constant temperature on pediatric patients intra-operatively3. We want to investigate the differences in temperature between the two approaches, covering and not covering pediatric patients, during induction of general anesthesia of a urologic procedure with a caudal block and the difference in temperature post-operatively. We hypothesize that the core temperatures of:

1. the covered and warmed group during induction of general anesthesia will be greater by 0.5ºC than the uncovered group during induction of general anesthesia.
2. both groups, covered and uncovered, will be equal during surgery and post-operatively. In other words, due to the active warming procedures during surgery and post-operatively in the PICU, core temperatures of the uncovered group will catch up to the covered group.

ELIGIBILITY:
Inclusion Criteria:

* The ages of the subjects ranging from 6 months to 3 years undergoing surgery for circumcision or hernia repair with caudal block.

Exclusion Criteria:

* ASA physical status classification greater than 2, unsigned or unattainable written informed consent form, induction of general anesthesia time of greater than 45 minutes, fever, or temperature regulation inability.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in an academic center
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Covered group during induction of general anesthesia will be greater by 0.5ºC than the uncovered group during induction of general anesthesia. | 1.5 years

SECONDARY OUTCOMES:
Covered and uncovered, will be equal during surgery and post-operatively. In other words, due to the active warming procedures during surgery and post-operatively in the PICU, core temperatures of the uncovered group will catch up to the covered group. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mohanad Shukry, MD, Principal Investigator — The University of Oklahoma Health Sciences Center
Locations (1):
- The University of Oklahoma Health Sciences Center Deparment of Anesthesiology, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Bissonnette B. Temperature monitoring in pediatric anesthesia. Int Anesthesiol Clin. 1992 Summer;30(3):63-76. PMID 1516974
- [Background] Hynson JM, Sessler DI, Moayeri A, McGuire J, Schroeder M. The effects of preinduction warming on temperature and blood pressure during propofol/nitrous oxide anesthesia. Anesthesiology. 1993 Aug;79(2):219-28, discussion 21A-22A. doi: 10.1097/00000542-199308000-00005. PMID 8342834